CLINICAL TRIAL: NCT05385016
Title: The Promotion of Healthy Lifestyles for Young Adults With Intellectual Disabilities
Brief Title: Cooking Classes for Young Adults With ID
Acronym: ChefBoyID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Study 148424
Record Dates: First submitted 2022-05-02; First posted 2022-05-23 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Intellectual Disability, Mild to Moderate
MeSH Terms: conditions — Intellectual Disability | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Education Arm (Experimental): Participants will attend weekly two hour small group instruction sessions. All sessions will have an education component, a hands-on nutrition/cooking lesson, and a group exercise session. Two health educators will be present during group sessions with one leading
  Interventions: Behavioral: Cooking Skills; Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Cooking Skills — This session will consist of a hands-on cooking demonstration in a demo kitchen. Skills addressed in this portion of the session will include proper kitchen utensil and appliance use, measuring dry and wet ingredients, following/reading a recipe, preparing ingredients, cooking a meal, etc. The participant will follow a visual recipe that provides a breakdown of each skill needed to complete each step of the recipe. Additionally, during the cooking session investigators will address nutrition topics related to food/kitchen safety, basic nutrition education (i.e., portion sizes, food groups, reading food labels, meal planning etc.) in a discussion format.
Behavioral: Physical Activity — This session will consist of a group functional fitness class. Each session will include a warm-up (~5 min) moderate-to-vigorous intensity aerobic and resistance exercise (~20 min) and cool-down/stretching (~5 min). Exercises may be accompanied by music and will include walking/jogging, dancing, imitating animal movements, vertical/horizontal jumps, squats, hurdles, walking on balance beam etc. Thera-Band, kettle bells, free weights, and medicine balls will be used during strength exercises for major muscle groups. These sessions will be led by certified personal trainers with experience in adaptive physical activity.

SUMMARY:
The purpose of this study is to examine the feasibility and initial efficacy of a healthy lifestyles intervention for the prevention of weight gain and the promotion of basic life skills related to improving health in transition age young adults with intellectual disabilities.

DETAILED DESCRIPTION:
This is a single arm, longitudinal trial. 30 young adults with intellectual disabilities will be recruited to participate in a 12-week, healthy lifestyles intervention, delivered in person to a group of individuals with ID at the Center for Children's Healthy Lifestyles and Nutrition. Participants will be asked to attend one 2 hr group session each week (~5-6 participants per group). All sessions will have an education component, a hands-on nutrition/cooking lesson, and a group exercise session. Additionally, participants will be asked to attend a 20-minute monthly individual goal setting session conducted remotely over Zoom video conferencing. All sessions will be conducted by a trained health educator experienced in working with individuals with intellectual disabilities. Tablet computers and Fitbit wireless activity monitors will be provided to all participants, with study issued HIPPA compliant Zoom and Fitbit accounts. Outcome assessments will be collected at baseline and after the 12-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an Intellectual Disability.
* Age: 18-30 yrs.
* Functional ability sufficient to understand directions and to communicate through spoken language.
* Reside in a supported living condition either at home or with no more than 1-4 residents and have a study partner (i.e., parent, staff who agrees to serve as support partner).
* Wireless Internet access in the home.
* Ability to walk without assistance.
* Consent from physician to do physical activity.

Exclusion Criteria:

* Actively participating in another research study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Attendance | Across 12 weeks
  The health coach will record attendance at all sessions. The outcome variable will be the percentage of attendance out of the total 12 scheduled exercise sessions attended.
Retention | Across 12 weeks
  We will calculate the percent of participants who complete the 12 week intervention.

SECONDARY OUTCOMES:
Cooking Skills | Change from Baseline to 12 weeks
  Cooking skills will be assessed by select questions from The Assessment of Functional Living Skills: Independent Living Skills. Parents/caregivers will fill this survey out on behalf of the participant.
Fitness | Change from Baseline to 12 weeks
  Fitness will be assessed using the 2 minute step test.
Lower Body Strength | Change from Baseline to 12 weeks
  Lower body muscle strength will be assessed using a standard 5-repetition maximum protocol on a Cybex plate-loaded leg press calculated with the Brzycki et al. 1-repetition maximum prediction equation. Grip strength will be measured using a hand dynamometer.
Upper Body Strength | Change from Baseline to 12 weeks
  Upper body strength will be assessed by grip strength, measured using a hand dynamometer.
Height | Change from Baseline to 12 weeks
  Standing height will be measured in duplicate with a portable stadiometer.
Weight | Change from Baseline to 12 weeks
  Participants will be weighed in duplicate, on a calibrated scale to the nearest 0.1 kg.
Waist circumference | Change from Baseline to 12 weeks
  Waist circumference will be assessed. Three measurements will be obtained with the outcome recorded as the average of the closest 2 measures.
Body Mass Index | Change from Baseline to 12 weeks
  Body Mass Index will be calculated as weight (kg)/height(m) squared.
Caregiver Stress | Change from Baseline to 12 weeks
  Caregiver stress will be assessed using the Parental Stress Scale. The Parental Stress Scale is an 18-item questionnaire assessing parents' feelings about their parenting role, exploring both positive aspects (e.g., emotional benefits, personal development, etc.) and negative aspects of parenthood (e.g., demands on resources, feelings of stress, etc.).Parental stress scores range from 18 to 90, with lower scores indicating lower levels of parental stress.
Accelerometer | Change from Baseline to 12 weeks.
  Physical activity will be assessed by accelerometer. Participants will be asked to wear the accelerometer around their waist for 7 days and than return in a pre-paid envelope
Daily Physical Activity | Across 12 weeks
  Daily physical activity across the 12 week study activity will be assessed using a Fitbit Versa 3 monitor worn on the non-dominant wrist during each day of the intervention
Individual Goals | Across 12 weeks
  Individual participant goals will be created and measured using The Goal Attainment Scale template during the individual education sessions. At least one physical activity goal and one nutrition goal will be measured per participant. The Goal Attainment Scale is an individualized outcome measure involving goal selection and goal scaling that is standardized in order to calculate the extent to which a participant's goals are met. Scores range from -2 to 2, which a higher scale indicating the most favorable outcome.
Work Capacity | Across 12 weeks
  Changes to fitness-related outcomes will be assessed by work capacity, once per month during the group exercise sessions. Performance will be evaluated based on the total number of rounds and repetitions (i.e., volume) of all movements completed during a 10-minute period (e.g., 3 rounds + 12 repetitions).

OTHER OUTCOMES:
Semi Structure Interview | Week 12
  Semi-structured interviews (audio recorded) will be conducted with the participant and their study partner following completion of the intervention to gather information on the overall ease and enjoyment of the program, changes in self-determination and healthy lifestyles, and suggestions to improve the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Danon JC, Koon L, Sherman JR, Rice AM, Quaife S, Helsel BC, Bodde A, Ptomey LT. Feasibility and preliminary efficacy of a skill-based lifestyle intervention for enhancing cooking abilities and physical fitness in young adults with intellectual disabilities. Disabil Health J. 2025 Apr;18(2):101767. doi: 10.1016/j.dhjo.2024.101767. Epub 2024 Dec 4. PMID 39648079